CLINICAL TRIAL: NCT05933005
Title: A Randomized, Double-blind, Parallel-group, Exploratory Clinical Trial to Evaluate Executive Function and Cognitive Improvement After Intervention Utilizing a Computerized Cognitive Rehabilitation Program (D-kit/EF1) in Children With Borderline Intellectual Functioning or Mild Intellectual Disability (FSIQ 50 - 85)
Brief Title: Intervention Utilizing a Computerized Cognitive Rehabilitation Program (D-kit/EF1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: DoBrain Inc. (Industry); Korea Health Industry Development Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-39462
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Mild Intellectual Disability; Borderline Intellectual Functioning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: This clinical trial is conducted using a double-blind design, requiring both the evaluators and participants to maintain blindness. The randomization table is prepared by an independent statistician who seals each copy of the randomization table separately after the allocation of the investigational device and control device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- D-kit/EF1 group (Experimental): The experimental group will use the D-kit/EF1 program on a mobile tablet device at least 5 times a week for 30 minutes each session, for a duration of 12 weeks.
  The program will be performed under the supervision of the participant's parents or primary caregivers, following the provided program usage guide.
  Interventions: Device: D-kit/EF1
- Sham group (Sham Comparator): The sham group will watch an educational animation video on a mobile tablet device at least 5 times a week for 30 minutes each session, for a duration of 12 weeks.
  The sham program was designed to provide a similar experience as the experimental group by replacing the content within the same app. The control group uses the same mobile tablet device and accesses the app with the provided control group account. When accessing the app with the control group account, instead of the Adaptive Learning Lesson reflecting the principles of D-kit, educational animations created for educational purposes are provided.
  The educational animations are original animations created by DOBAIN Inc..
  Interventions: Device: Sham group program

INTERVENTIONS:
Device: D-kit/EF1 — D-kit/EF1 delivers interventions through online platforms and can be downloaded to smart devices through the iOS App store or Google Play Store. Games are specifically designed to assist children with delayed cognitive development in the acquisition of foundational cognitive skills.
  The core technology of the D-kit/EF1 is the 'reinforcement technique', a technology used in traditional behavioral therapy. Specifically, D-kit incorporates the Discrete Trial Training (DTT) approach into its instructional content to facilitate the acquisition of basic cognitive skills.
  Arms: D-kit/EF1 group
Device: Sham group program — The sham program was designed to provide a similar experience as the experimental group by replacing the content within the same app. The control group uses the same mobile tablet device and accesses the app with the provided control group account. When accessing the app with the control group account, instead of the Adaptive Learning Lesson reflecting the principles of D-kit, educational animations created for educational purposes are provided.
  Arms: Sham group

SUMMARY:
The goal of this exploratory clinical trial is to test the effects of the computerized cognitive rehabilitation program (D-kit/EF1) for children with borderline intellectual functioning or mild intellectual disability after its use.

Participants will use the D-kit/EF1 program on an iOS device 5 times a week for 30 minutes each session, for a duration of 12 weeks.

Researchers will compare treatment group that uses D-kit/EF1 with sham group that watches educational videos on the same iOS device.

DETAILED DESCRIPTION:
This clinical trial is a randomized, double-blind, parallel-group, exploratory study to confirm the efficacy of a computerized cognitive rehabilitation program (D-kit/EF1) in cognitive improvement of children with borderline intellectual functioning or mild intellectual disability (FSIQ 50 - 85).

D-kit/EF1, a computerized cognitive rehabilitation program, incorporates game-type quizzes to enhance executive function in children with Mild Intellectual Disability (MID) or Borderline Intellectual Functioning (BIF) as an adjunctive treatment alongside the current standard of care (SOC). D-kit/EF1 delivers interventions through online platforms and can be downloaded to smart devices through the iOS App store or Google Play Store. Games are specifically designed to assist children with delayed cognitive development in the acquisition of foundational cognitive skills.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4-8 years (48-96 months) of both genders at the time of obtaining consent.
2. Children with borderline intellectual functioning or mild intellectual disability (FSIQ 50-85) who meet the following criteria within 3 months of screening:

   * Stanford-Binet Intelligence Scale - 5th edition (SB-5) criteria: FSIQ 50-85.
   * NIH Toolbox Cognition Battery (NIHTB-CB) DCCS score of 7 or lower.
3. Children who are capable of communicating and behaving at a level sufficient to participate in the required tests and therapeutic activities of this clinical trial.
4. Individuals for whom the legal guardian and primary caregiver have voluntarily decided to participate in this clinical trial after receiving sufficient explanation and have provided written consent to comply with the requirements of the clinical trial.

Exclusion Criteria:

1. If the parents or primary caregiver of the trial subjects, who will perform the key assessments on the trial subjects, are unable to read or write in English, thus are impossible to conduct the assessments.
2. Patients with conditions (e.g., blindness, color blindness, hearing loss, or deafness) that make it difficult to perform the digital therapy of the medical device for the clinical trial, D-kit/EF1, and the key assessment item for the clinical trial, NIHTB-CB DCCS test.
3. If the subject has participated in another clinical trial or has been administered investigational drugs for clinical trial purposes within the 4 weeks prior to screening (except, cases where the subject has not received investigational drugs or has participated in non-interventional observational studies are eligible for enrollment).
4. Other subjects who are deemed unsuitable for participation in this clinical trial based on the judgment of the investigators.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in NIHTB-CB DCCS Computed Score from Baseline to Week 12 | Baseline (Week 0), Post-treatment (Week 12)
  DCCS is assessed to evaluate the subjects' executive function and cognitive function. Two target pictures that differ across two dimensions are presented to the participants. Participants are asked to match a series of bivalent test pictures to target pictures, first according to one dimension, and after a number of trials, according to the other dimension. "Switch" trials are also employed, in which the participants must change the dimension. Scoring is based on a combination of accuracy and reaction time. A 2-vector scoring method is employed that uses accuracy and reaction time, where each of these "vectors" ranges in value between 0 and 5, and the computed score, combining each vector score, ranges in value from 0 - 10. 95% confidence interval of the mean difference for the change in scores will be calculated. To test for differences in DCCS Computed scores change, either a two-sample t-test or Wilcoxon's rank sum test will be used, depending on the normality assumption.

SECONDARY OUTCOMES:
Change in NIHTB-CB DCCS Computed Score from Baseline to Week 16 | Baseline (Week 0), Follow-up (Week 16)
  DCCS is assessed to evaluate the subjects' executive function and cognitive function. Two target pictures that differ across two dimensions are presented to the participants. Participants are asked to match a series of bivalent test pictures to target pictures, first according to one dimension, and after a number of trials, according to the other dimension. "Switch" trials are also employed, in which the participants must change the dimension. Scoring is based on a combination of accuracy and reaction time. A 2-vector scoring method is employed that uses accuracy and reaction time, where each of these "vectors" ranges in value between 0 and 5, and the computed score, combining each vector score, ranges in value from 0 - 10. 95% confidence interval of the mean difference for the change in scores will be calculated. To test for differences in DCCS Computed scores change, either a two-sample t-test or Wilcoxon's rank sum test will be used, depending on the normality assumption.
Change in Vineland-3 Score from Baseline to Week 12 | Baseline (Week 0), Post-treatment (Week 12)
  The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) is a parent interview that measures a child's everyday adaptive skills at home and in the community in the areas of: Communication, Daily Living Skills, Socialization, and Motor. Each domain and the overall Adaptive Behavior Composite (ABC) result in a norm-referenced standard score. The domain scores are also expressed as standard scores with a mean of 100 and standard deviation of 15. Individuals with domain and ABC Standard Scores of 130 to 140 are considered to have a high adaptive level, 115 to 129 is considered moderately high, 86 to 114 as adequate, 71 to 85 as moderately low and 20 to 70 as low.
Change in Vineland-3 Score from Baseline to Week 16 | Baseline (Week 0), Follow-up (Week 16)
  The Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) is a parent interview that measures a child's everyday adaptive skills at home and in the community in the areas of: Communication, Daily Living Skills, Socialization, and Motor. Each domain and the overall Adaptive Behavior Composite (ABC) result in a norm-referenced standard score. The domain scores are also expressed as standard scores with a mean of 100 and standard deviation of 15. Individuals with domain and ABC Standard Scores of 130 to 140 are considered to have a high adaptive level, 115 to 129 is considered moderately high, 86 to 114 as adequate, 71 to 85 as moderately low and 20 to 70 as low.
Change in BRIEF-P or BRIEF-2 Global Executive Composite Score from Baseline to Week 12 | Baseline (Week 0), Post-treatment (Week 12)
  Behavior Rating Inventory of Executive Function Preschool (BRIEF-P) and Behavior Rating Inventory of Executive Function, 2nd Edition (BRIEF-2) measure multiple aspects of executive functioning. BRIEF-P is administered for children aged 4 at point of evaluation, and BRIEF-2 is administered for children aged 5 or older at point of evaluation. T scores are used to interpret the child's level of executive functioning on the BRIEF-P and BRIEF-2. T scores from 60 to 64 are considered mildly elevated, and T scores from 65 to 69 are considered potentially clinically elevated. T scores at or above 70 are considered clinically elevated.
Change in BRIEF-P or BRIEF-2 Global Executive Composite Score from Baseline to Week 16 | Baseline (Week 0), Follow-up (Week 16)
  Behavior Rating Inventory of Executive Function Preschool (BRIEF-P) and Behavior Rating Inventory of Executive Function, 2nd Edition (BRIEF-2) measure multiple aspects of executive functioning. BRIEF-P is administered for children aged 4 at point of evaluation, and BRIEF-2 is administered for children aged 5 or older at point of evaluation. T scores are used to interpret the child's level of executive functioning on the BRIEF-P and BRIEF-2. T scores from 60 to 64 are considered mildly elevated, and T scores from 65 to 69 are considered potentially clinically elevated. T scores at or above 70 are considered clinically elevated.

CONTACTS AND LOCATIONS:
Overall Officials: Young Shin Kim, MD PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Nancy Friend Pritzker Psychiatry Building, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No